CLINICAL TRIAL: NCT05481606
Title: Clinical Outcomes of Cesarean Scar Pregnancy With Different Type: a Prospective Cohort Study
Brief Title: Cesarean Scar Pregnancy and Clinical Outcomes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Zhao Yangyu, Chief of obstetrics, Peking University Third Hospital
Other Study IDs: PKUTH22-07-27
Record Dates: First submitted 2022-07-27; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Blood Loss; Repeat Cesarean Section; Maternal Transmission; Hysterectomy; Placenta Accreta Spectrum; Abortion
MeSH Terms: conditions — Hemorrhage; Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — hair, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type I: 1) the gestational sac is partially implanted in the uterine scar, partially or mostly located in the uterine cavity, and a few may even reach the uterine cavity at the bottom of the palace; 2) the gestational sac is significantly deformed, and elongated, and its the lower end presented a acute Angle; 3) The myometrium between the gestational sac and the bladder became thinner, with a thickness of >3 mm; 4) Doppler flow image: trophoblast blood flow signal can be seen in the scar (low resistance blood flow)
- Type II: 1) The gestating sac is partially implanted in the scar of the uterus, partially or mostly located in the uterine cavity, and a few may even reach the uterine cavity at the bottom of the uterus; 2)the gestational sac is significantly deformed, and elongated, and its the lower end presented a acute Angle; 3) The myometrium between the stretch and the bladder becomes thinner (3 mm in thickness); 4) color Doppler flow image: trophoblast blood flow signal (low resistance blood flow) can be seen in the scar.
- Type III: 1) The gestating sac is completely implanted in the muscle layer of the scar of the uterus and protrudes outward toward the bladder; 2) Uterine cavity and cervical canal emptiness; 3) The myometrium between the gestational sac and the bladder was significantly thinner or absent, with a thickness of 3 mm; 4) color Doppler flow image: trophoblast blood flow signal (low resistance blood flow) can be seen in the scar. Among them, there is a special ultrasonic manifestation of cesarean scar pregnancy in type III, namely mass type, whose sonographic characteristics

SUMMARY:
This study is a prospective cohort study, led by Prof. Zhao Yangyu, from the Department of Gynecology & Obstetrics, Peking University Third Hospital.

DETAILED DESCRIPTION:
Cesarean section, myomectomy and other surgeries for uterus are likely to cause scars in different parts of the uterus. During the subsequent pregnancy, the incidence rate of cesarean scar pregnancy, placenta previa, placenta increta and the risk of termination of the first and mid-trimester pregnancy is likely to increase. Cesarean scar pregnancy is regarded as a risk factor of uterine rupture in the third trimester of pregnancy or delivery period, which severely affects the maternal and perinatal health and safety. This study is planning to prospectively include pregnant women aged 20-49 years from Peking University Third Hospital. All women with diagnosis on cesarean scar pregnancy was included prior to 14 wks of gestation. We divided the women into three different groups: type I, type II and type III according to characteristics in gestation sac,uterine scar, bladder, the latter with potentially worse outcomes in term of maternal morbidity and mortality. Data including demographics, medical history, reproductive history, prenatal health care, gestational complications, and pregnancy and birth outcomes will be collected via electronic data capture system.

ELIGIBILITY:
Inclusion Criteria:

* Female aged ≥ 20 years
* Female with cesarean scar pregnancy
* Less than 14 gestational weeks
* Planning to receive prenatal healthcare and delivery service at the study hospital

Exclusion Criteria:

* Inability to provide informed consent
* Women with mental disorders

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study is planning to include 1000 pregnant women with uterine scar aged 20 years from Peking University Third Hospital. Pregnant women who are planning to recieve prenatal healthcare and delivery in this hospital are potential candidates for the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of blood loss | delivery
  blood loss
Incidence of postpartum hemorrhage | delivery
  postpartum hemorrhage
Incidence of maternal transfusion | delivery
  maternal transfusion
Incidence of spontaneous abortion | delivery
  spontaneous abortion
Incidence of stillbirth | delivery
  stillbirth
Incidence of perinatal death | 42 days postpartum
  perinatal death

SECONDARY OUTCOMES:
Maternal death | At 24-28 weeks
  Deaths during pregnancy or less than 42 days after termination of pregnancy
Maternal death | 42 days postpartum
  Deaths during pregnancy or less than 42 days after termination of pregnancy
The rate of repeated cesarean delivery | At delivery
  Cesarean rate is defined as the number of cesarean delivery divided by the number of live births.

IPD SHARING:
Plan to Share IPD: Undecided